CLINICAL TRIAL: NCT05948254
Title: Utilized Scan Body Technique For Jaw Relation Registration And Face Scan Alignment (Triple Function Scan Body)
Brief Title: Utilized Scan Body Technique For Triple Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 245862
Record Dates: First submitted 2023-07-10; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2022-05

CONDITIONS: Digital Technology; Dental Implant; Occlusion
Keywords: Jaw relation; Scan body; Full arch dental implants
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Intervention Model Description: Triple Function Scan Body
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Triple Function Scan Body (Other): Full arch implants were placed, a triple function scan Body and thus simplifying the workflow for full arch cases and reducing the number of visits to only 3 visits. Scan bodies were utilized for implant position scanning, facial scan alignment and as stoppers for jaw relation capturing as scan bodies were used as stoppers for jaw relation registration.
  Interventions: Procedure: Triple function scan body

INTERVENTIONS:
Procedure: Triple function scan body — The scan bodies were used to scan the implant position, Jaw registration and facial scan alignment, First of all scan bodies were selected according to vertical dimension of occlusion, then the emergence profile together with the selected scan body were scanned,All scan bodies were then removed from the patient mouth except one or even two that were scanned in the jaw scan step, this scan body was utilized as a stopper, the patient was asked to bite until the scan body came in contact with the lower or upper teeth in case of edentulous upper or lower arch respectively, scan body in place (in the same orientation of the previous jaw scan ) provided that at least the tip of the scan body appeared when the patient is asked to smile which would be used as a common area so that the intra oral scanner can relate the jaw scan to the lips and face.

SUMMARY:
A triple function scan Body were done on healed dental implant, thus simplifying the workflow for full arch cases and reducing the number of visits to only 3 visits. In this technique, scan bodies were utilized for implant position scanning, facial scan alignment and as stoppers for jaw relation capturing as scan bodies were used as stoppers for jaw relation registration.

DETAILED DESCRIPTION:
The present article describes a novel technique for merging a patient's facial scan with implant scan body and in the same time utilizing the same scan body for recording the jaw relation in only one visit. As a result, a facially driven full-arch implant-supported interim prosthesis can be fabricated first followed by the final restoration in a simplified approach. The aim of this study is to determine whether there is a difference between virtual design and reality using scan body technique (triple function scan body which reflects the accuracy of the scanning protocol. The null hypothesis established that there was consistency between the virtual design and prosthesis in patient's mouth. The scan body was placed in the edentulous arch in the jaw scan step so that bite registration would be easier for the intraoral scanner (IOS) in order to be able to capture both the teeth of the antagonist and part of the scan body in the edentulous jaw simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* patient had at least one edentulous arch with at least 5 osseointegrated implants with healing period of 3 months after surgical procedure.
* Implants are stable
* Systemically free

Exclusion Criteria:

* Smokers
* Uncooperative patients

Ages: 22 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
percentage of consistency in simultaneous contacts in maximal intercuspal position | 2 months following the final prosthesis
  At 2 months follow up after final prostheses delivery, a frontal photo was taken and an intra oral scan was made for each patient in order to assess the degree of consistency between initial virtual design and reality using Exocad Software, The intra oral Scan of the full arch restoration is inserted into Exocad Software and the interocclusal contacts for all teeth were detected, classifying them in a dichotomy variable (yes/no) contact or not per tooth.

CONTACTS AND LOCATIONS:
Overall Officials: Doaa Adel-Khattab, PhD, Principal Investigator — Associate Professor Faculty of Dentistry, Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Abbassia, Egypt

IPD SHARING:
Plan to Share IPD: No